CLINICAL TRIAL: NCT02165397
Title: iNNOVATE Study: A Randomized, Double-Blind, Placebo- Controlled, Phase 3 Study of Ibrutinib or Placebo in Combination With Rituximab in Subjects With Waldenström's Macroglobulinemia
Brief Title: Ibrutinib With Rituximab in Adults With Waldenström's Macroglobulinemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacyclics LLC. (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PCYC-1127-CA
Record Dates: First submitted 2014-06-09; First posted 2014-06-17 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2020-12

CONDITIONS: Waldenström's Macroglobulinemia
Keywords: Ibrutinib; Pharmacyclics; PCYC; Lymphoma; Btk inhibitor; WM; Rituximab; Rituxan; Waldenström's; Waldenstrom Macroglobulinemia; non-Hodgkin lymphoma; NHL
MeSH Terms: conditions — Waldenstrom Macroglobulinemia; Lymphoma; Lymphoma, Non-Hodgkin | interventions — ibrutinib; Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Randomized Study (Ibrutinib + Rituximab) (Experimental): Ibrutinib: 420 mg (3 capsules x 140 mg) orally administered daily beginning from Day 1. Rituximab: 375 mg/m^2 intravenous (IV) per package insert weekly for four consecutive weeks, followed by a second four-weekly rituximab course after a three-month interval.
  Interventions: Drug: Ibrutinib; Drug: Rituximab
- Randomized Study (Placebo + Rituximab) (Experimental): Placebo: 3 capsules of placebo orally administered daily beginning from Day 1. Rituximab: 375 mg/m^2 IV per package insert weekly for four consecutive weeks, followed by a second four-weekly rituximab course after a three-month interval.
  Interventions: Drug: Placebo; Drug: Rituximab
- Open-Label Substudy (Ibrutinib) (Experimental): Ibrutinib: 420 mg (3 capsules) orally administered daily beginning from Day 1.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Participants will receive 420 mg of Ibrutinib orally.
  Other Names: PCI-32765
  Arms: Open-Label Substudy (Ibrutinib); Randomized Study (Ibrutinib + Rituximab)
Drug: Placebo — Participants will receive placebo capsules orally.
  Arms: Randomized Study (Placebo + Rituximab)
Drug: Rituximab — Participants will receive rituximab 375 mg/m^2 IV.
  Other Names: Rituxan
  Arms: Randomized Study (Ibrutinib + Rituximab); Randomized Study (Placebo + Rituximab)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ibrutinib in combination with rituximab in participants with Waldenström's macroglobulinemia (WM).

ELIGIBILITY:
Eligibility Criteria for the Randomized Study

Inclusion Criteria:

* Untreated or previously treated for WM. Previously treated subjects must have either documented disease progression or had no response (stable disease) to the most recent treatment regimen
* Centrally confirmed clinicopathological diagnosis of WM
* Measurable disease defined as serum monoclonal immunoglobulin M (IgM) >0.5 g/dL
* Symptomatic disease meeting at least 1 of the recommendations from the Second International Workshop on Waldenström Macroglobulinemia for requiring treatment
* Hematology and biochemical values within protocol-defined limits
* Men and women ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2

Exclusion Criteria:

* Known involvement of the central nervous system by WM
* Disease that is refractory to the last prior rituximab-containing therapy defined as either

  * Relapse after the last rituximab-containing therapy < 12 months since last dose of rituximab, OR
  * Failure to achieve at least a minor response (MR) after the last rituximab-containing therapy If the subject meets this exclusion criterion and therefore is excluded from the main randomized study, participation in the non randomized substudy (Arm C) may be considered
* Rituximab treatment within the last 12 months before the first dose of study drug
* Known anaphylaxis or (immunoglobulin E) IgE-mediated hypersensitivity to murine proteins or to any component of rituximab
* Prior exposure to ibrutinib or other Bruton's tyrosine kinase (BTK) inhibitors
* Known bleeding disorders (eg, von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 12 months prior to enrollment.
* Any uncontrolled active systemic infection.
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
* Currently active, clinically significant cardiovascular disease
* Requires treatment with a strong cytochrome P450 (CYP) 3A inhibitor

Eligibility Criteria for Open-label Substudy Treatment Arm C

The inclusion/exclusion criteria for the substudy (Arm C) are identical to those described above for the randomized study but, to be eligible, subjects need to be considered refractory to the last prior rituximab-containing therapy defined as either

* Relapse after the last rituximab-containing therapy <12 months since last dose of rituximab, OR
* Failure to achieve at least a MR after the last rituximab-containing therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2019-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernhard Hauns, MD, Study Director — Pharmacyclics LLC.
Locations (48):
- United States (10):
  - University of California Los Angeles, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Australia (4):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Concord Repartriation General Hospital, Concord, New South Wales
  - Flinders Medical Center, Bedford Park, South Australia
  - Peter MacCallum Cancer Center, Melbourne, Victoria
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Queen Elizabeth II Health Sciences Center, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
- France (10):
  - Institut Paoli-Calmettes, Marseille, Bouches-du-Rhône
  - Centre Hospitalier de Saint Brieuc Hopital Yves le Foll, Saint-Brieuc, Finistère
  - Hôtel Dieu, Nantes, Loire-Atlantique
  - CHU de Nancy-Hopital Brabois Adulte, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hôpital Claude Huriez, Lille, Nord
  - CHU Estaing, Clermont-Ferrand, Puy-de-Dôme
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhône
  - Hopital Henri Mondor, Créteil
  - Hôpital Saint Louis, Paris
  - Groupe Hospitalier Pitié Salpétrière, Paris
- Germany (5):
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen, Baden-Wurttemberg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Universität Des Saarlandes, Homburg, Saarland
  - DIAKO Evangelische Diakonie Krankenhaus gGmbH, Bremen
  - LMU Klinikum der Universität München, München
- Greece (4):
  - University General Hospital of Patras, Pátrai, Achaia
  - Alexandra Hospital, Athens, Attica
  - University General Hospital of Thessaloniki "AHEPA", Thessaloniki, Macedonia
  - Laiko General Hospital of Athens, Athens
- Italy (5):
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - ASST di Pavia - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - Azienda Ospedaliero Universitaria Santa Maria della Misericordia di Udine, Udine
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Salamanca, Salamanca, Castille and León
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Infanta Leonor, Madrid
- Royal Bournemouth Hospital, Bournemouth, Dorset, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Requests for access to individual participant data from clinical studies conducted by Pharmacyclics LLC, an AbbVie Company, can be submitted through Yale Open Data Access (YODA) Project site at the following link.
URL: http://yoda.yale.edu

REFERENCES:
- [Background] Dimopoulos MA, Tedeschi A, Trotman J, Garcia-Sanz R, Macdonald D, Leblond V, Mahe B, Herbaux C, Tam C, Orsucci L, Palomba ML, Matous JV, Shustik C, Kastritis E, Treon SP, Li J, Salman Z, Graef T, Buske C; iNNOVATE Study Group and the European Consortium for Waldenstrom's Macroglobulinemia. Phase 3 Trial of Ibrutinib plus Rituximab in Waldenstrom's Macroglobulinemia. N Engl J Med. 2018 Jun 21;378(25):2399-2410. doi: 10.1056/NEJMoa1802917. Epub 2018 Jun 1. PMID 29856685
- [Background] Dimopoulos MA, Trotman J, Tedeschi A, Matous JV, Macdonald D, Tam C, Tournilhac O, Ma S, Oriol A, Heffner LT, Shustik C, Garcia-Sanz R, Cornell RF, de Larrea CF, Castillo JJ, Granell M, Kyrtsonis MC, Leblond V, Symeonidis A, Kastritis E, Singh P, Li J, Graef T, Bilotti E, Treon S, Buske C; iNNOVATE Study Group and the European Consortium for Waldenstrom's Macroglobulinemia. Ibrutinib for patients with rituximab-refractory Waldenstrom's macroglobulinaemia (iNNOVATE): an open-label substudy of an international, multicentre, phase 3 trial. Lancet Oncol. 2017 Feb;18(2):241-250. doi: 10.1016/S1470-2045(16)30632-5. Epub 2016 Dec 10. PMID 27956157
- [Derived] Guijosa A, Ramirez-Gamero A, Sarosiek S, Branagan AR, von Keudell G, Treon SP, Castillo JJ. Ibrutinib plus rituximab vs ibrutinib monotherapy in patients with Waldenstrom macroglobulinemia: a pooled analysis. Blood Adv. 2025 Sep 23;9(18):4705-4715. doi: 10.1182/bloodadvances.2025016536. PMID 40674744
- [Derived] Buske C, Tedeschi A, Trotman J, Garcia-Sanz R, MacDonald D, Leblond V, Mahe B, Herbaux C, Matous JV, Tam CS, Heffner LT, Varettoni M, Palomba ML, Shustik C, Kastritis E, Treon SP, Ping J, Hauns B, Arango-Hisijara I, Dimopoulos MA. Plain Language Summary of the iNNOVATE study: ibrutinib plus rituximab is well-tolerated and effective in people with Waldenstrom's macroglobulinemia. Future Oncol. 2023 Feb;19(5):345-353. doi: 10.2217/fon-2022-1015. Epub 2023 Feb 23. PMID 36815271
- [Derived] Buske C, Tedeschi A, Trotman J, Garcia-Sanz R, MacDonald D, Leblond V, Mahe B, Herbaux C, Matous JV, Tam CS, Heffner LT, Varettoni M, Palomba ML, Shustik C, Kastritis E, Treon SP, Ping J, Hauns B, Arango-Hisijara I, Dimopoulos MA. Ibrutinib Plus Rituximab Versus Placebo Plus Rituximab for Waldenstrom's Macroglobulinemia: Final Analysis From the Randomized Phase III iNNOVATE Study. J Clin Oncol. 2022 Jan 1;40(1):52-62. doi: 10.1200/JCO.21.00838. Epub 2021 Oct 4. PMID 34606378
- [Derived] Trotman J, Buske C, Tedeschi A, Matous JV, MacDonald D, Tam CS, Tournilhac O, Ma S, Treon SP, Oriol A, Ping J, Briso EM, Arango-Hisijara I, Dimopoulos MA. Single-Agent Ibrutinib for Rituximab-Refractory Waldenstrom Macroglobulinemia: Final Analysis of the Substudy of the Phase III InnovateTM Trial. Clin Cancer Res. 2021 Nov 1;27(21):5793-5800. doi: 10.1158/1078-0432.CCR-21-1497. Epub 2021 Aug 11. PMID 34380643

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 48 sites (10 in the United States, 30 in Europe, 4 in Canada and 4 in Australia).
Pre-assignment Details: Participants were randomized in a 1:1 ratio to receive ibrutinib + rituximab (Ibr+R) or placebo + rituximab (Pbo+R). Separately, participants refractory to treatment with rituximab were enrolled in an open-label ibrutinib monotherapy substudy to further investigate the safety and efficacy of ibrutinib.
Groups:
- Ibrutinib + Rituximab: Ibrutinib: 420 mg (3 capsules) orally administered daily beginning from Day 1 in Week 1 until progression, discontinuation due to toxicity or other reasons to discontinue treatment.
  Rituximab: 375 mg/m^2 intravenous (IV) per package insert weekly for four consecutive weeks (Day 1 of Weeks 1-4), followed by a second four-weekly rituximab course after a three-month interval (Weeks 17-20) for a total of 8 infusions of rituximab.
- Placebo + Rituximab: Placebo: 3 capsules of placebo orally administered daily beginning from Day 1 in Week 1 until progression, discontinuation due to toxicity or other reasons to discontinue treatment.
  Rituximab: 375 mg/m^2 IV per package insert weekly for four consecutive weeks (Day 1 of Weeks 1-4), followed by a second four-weekly rituximab course after a three-month interval (Weeks 17-20) for a total of 8 infusions of rituximab.
- Open-Label Substudy: Ibrutinib: Ibrutinib: 420 mg (3 capsules) orally administered daily beginning from Day 1 in Week 1 until progression, discontinuation due to toxicity or other reasons to discontinue treatment. Participants (rituximab refractory) were treated in an open-label substudy independently of the 2 randomized main treatment arms.
Period: Overall Study
Arm/Group | Ibrutinib + Rituximab | Placebo + Rituximab | Open-Label Substudy: Ibrutinib
Started | 75 | 75 | 31
Completed (On-study until study termination by sponsor.) | 61 | 56 | 21
Not Completed | 14 | 19 | 10
Not completed — Death | 7 | 10 | 8
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Withdrawal by Subject | 6 | 6 | 1
Not completed — Other, Not Specified | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ibrutinib + Rituximab: Ibrutinib: 420 mg (3 capsules) orally administered daily beginning from Day 1 in Week 1 until progression, discontinuation due to toxicity or other reasons to discontinue treatment.
  Rituximab: 375 mg/m^2 IV per package insert weekly for four consecutive weeks (Day 1 of Weeks 1-4), followed by a second four-weekly rituximab course after a three-month interval (Weeks 17-20) for a total of 8 infusions of rituximab.
- Total: Total of all reporting groups
Arm/Group | Ibrutinib + Rituximab | Placebo + Rituximab | Open-Label Substudy: Ibrutinib | Total
Number analyzed (Participants) | 75 | 75 | 31 | 181
Age, Customized [Count of Participants; unit: Participants]
  < 65 years old | 28 | 30 | 14 | 72
  >= 65 years old | 47 | 45 | 17 | 109
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 21 | 11 | 62
  Male | 45 | 54 | 20 | 119
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 5
  Not Hispanic or Latino | 72 | 74 | 30 | 176
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 0 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 2
  White | 58 | 60 | 26 | 144
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 13 | 14 | 3 | 30

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Based on Independent Review Committee (IRC) Assessment - Kaplan Meier Landmark Estimates at Month 54
Description: PFS was defined as the time from date randomization to date of first IRC-confirmed disease progression (PD) assessed according to the modified VIth International Workshop on Waldenström's Macroglobulinemia (IWWM) criteria (National Comprehensive Cancer Network [NCCN] 2014) or death due to any cause, whichever occurs first, regardless of the use of subsequent antineoplastic therapy prior to documented PD or death.
  As the median PFS was not reached in the Ibrutinib + Rituximab arm at the time of the analysis, Kaplan Meier landmark estimate of the PFS rate at 54 months (that is, the estimated percentage of participants with PFS at Month 54) is presented.
Time Frame: Month 54 (median time on study: 49.7 months [Ibr+R and Pbo+R] and 57.9 months [Open-Label Ibr])
Population: Intent to Treat population: all randomized/enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibrutinib + Rituximab | Placebo + Rituximab | Open-Label Substudy: Ibrutinib
Number analyzed (Participants) | 75 | 75 | 31
percentage of participants | 68.0 [54.8 to 78.1] | 25.3 [15.3 to 36.6] | 39.7 [22.3 to 56.7]
Statistical Analysis 1: Comparison: Ibrutinib + Rituximab vs Placebo + Rituximab; Test type: Superiority; p < 0.0001, Log Rank — The treatment effect was tested with a stratified log rank test; Hazard Ratio (HR) = 0.250, 95% CI 2-sided [0.148 to 0.420] — The hazard ratio and its 95% confidence interval were based on a Cox regression model stratified by the randomization stratification factors

2. Secondary Outcome: Overall Response Rate (ORR) Based on IRC Assessment Up to 3 Years After Last Participant Randomized
Description: ORR, defined as the percentage of participants achieving a best overall response of protocol-specified complete response (CR), very good partial response (VGPR), or partial response (PR) per the IRC assessment at or prior to initiation of subsequent antineoplastic therapy and confirmed by 2 consecutive assessments. IRC assessment of response was conducted according to the modified VIth IWWM (NCCN 2014) criteria and incorporated assessments from the central radiology review. CR required complete resolution of lymphadenopathy/splenomegaly if present at baseline. VGPR and PR required reduction in lymphadenopathy/splenomegaly if present at baseline.. Kaplan-Meier estimate.
Time Frame: Median time on study: 49.7 months (Ibr+R and Pbo+R) and 57.9 months (Open-Label Ibr)
Population: Intent to Treat population: all randomized/enrolled participants
Measure: Number; unit: percentage of participants
Groups:
- Ibrutinib + Rituximab: Ibrutinib: 420 mg (3 capsules) orally administered daily beginning from Day 1 in Week 1 until progression, discontinuation due to toxicity or other reasons to discontinue treatment.
  Rituximab: 375 mg/m2 IV per package insert weekly for four consecutive weeks (Day 1 of Weeks 1-4), followed by a second four-weekly rituximab course after a three-month interval (Weeks 17-20) for a total of 8 infusions of rituximab.
- Placebo + Rituximab: Placebo: 3 capsules of placebo orally administered daily beginning from Day 1 in Week 1 until progression, discontinuation due to toxicity or other reasons to discontinue treatment.
  Rituximab: 375 mg/m2 IV per package insert weekly for four consecutive weeks (Day 1 of Weeks 1-4), followed by a second four-weekly rituximab course after a three-month interval (Weeks 17-20) for a total of 8 infusions of rituximab.
Arm/Group | Ibrutinib + Rituximab | Placebo + Rituximab | Open-Label Substudy: Ibrutinib
Number analyzed (Participants) | 75 | 75 | 31
percentage of participants | 76.0 | 30.7 | 77.4
Statistical Analysis 1: Comparison: Ibrutinib + Rituximab vs Placebo + Rituximab; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Response rate was compared using Cochran-Mantel-Haenszel (CMH) chi-square test; Rate Ratio = 2.526, 95% CI 2-sided [1.753 to 3.639]

3. Secondary Outcome: Time to Next Treatment (TnT) Time From the Date of Randomization to the Start Date of Any Subsequent WM Treatment.
Description: TTnT was measured from the date of randomization to the start date of any subsequent WM treatment. Participants without subsequent treatment were censored at the date of the last study visit.
  As the median TTnT was not reached in the Ibrutinib + Rituximab arm and the Open-Label Substudy arm at the time of the analysis, Kaplan Meier landmark estimate of the TTnT rate at 54 months (that is, the estimated percentage of participants not receiving subsequent WM treatment at Month 54) are presented.
Time Frame: Month 54 (median time on study: 49.7 months [Ibr+R and Pbo+R] and 57.9 months [Open-Label Ibr])
Population: Intent to Treat population: all randomized/enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibrutinib + Rituximab | Placebo + Rituximab | Open-Label Substudy: Ibrutinib
Number analyzed (Participants) | 75 | 75 | 31
percentage of participants | 87.4 [77.2 to 93.3] | 29.4 [18.2 to 41.6] | 64.6 [44.1 to 79.2]
Statistical Analysis 1: Comparison: Ibrutinib + Rituximab vs Placebo + Rituximab; Test type: Superiority; p < 0.0001, Log Rank — P-value is from a stratified log-rank test; Hazard Ratio (HR) = 0.102, 95% CI 2-sided [0.049 to 0.212] — Hazard ratio is estimated using a stratified Cox regression model

4. Secondary Outcome: Percentage of Participants With Sustained Hemoglobin (Hgb) Improvement Up to 3 Years After Last Participant Randomized
Description: Percentage of participants achieving a sustained improvement in Hgb at or prior to initiation of subsequent antineoplastic therapy. Hgb improvement is defined as an increase of ≥ 2 g/dL over baseline regardless of baseline value, or an increase to >11 g/dL with a ≥0.5 g/dL improvement if baseline is ≤ 11 g/dL. Sustained Hgb improvement is defined as improvement that is sustained continuously for ≥ 56 days (8 weeks) without blood transfusion or growth factors, which includes hemoglobin > 110 g/L with at least a 5 g/L improvement if baseline ≤110 g/L or increase ≥20 g/L over baseline.
Time Frame: Median time on study: 49.7 months (Ibr+R and Pbo+R) and 57.9 months (Open-Label Ibr)
Population: Intent to Treat population: all randomized/enrolled participants
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib + Rituximab | Placebo + Rituximab | Open-Label Substudy: Ibrutinib
Number analyzed (Participants) | 75 | 75 | 31
percentage of participants | 77.3 | 42.7 | 71.0
Statistical Analysis 1: Comparison: Ibrutinib + Rituximab vs Placebo + Rituximab; Test type: Superiority; p < 0.0001, Chi-squared; Rate Ratio = 1.813, 95% CI 2-sided [1.357 to 2.421]

5. Secondary Outcome: Percentage of Participants With ≥ 3 Points Increase From Baseline by Week 25 in the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Subscale Score
Description: Percentage of participants with ≥ 3 points increase from baseline by Week 25 in the FACIT-Fatigue subscale score.The FACIT-Fatigue is a 13-item questionnaire that assesses participant reported fatigue and its impact upon daily activities and function over the past 7 days. Each of the 13 items of the FACIT-Fatigue Scale ranges from 0-4, with a range of possible total scores from 0 (extreme fatigue) to 52 (no fatigue). Scores below 30 indicate severe fatigue.
Time Frame: Baseline, 25 weeks
Population: Intent to Treat population: all randomized/enrolled participants
Measure: Number; unit: percentage of participants
Arm/Group | Ibrutinib + Rituximab | Placebo + Rituximab | Open-Label Substudy: Ibrutinib
Number analyzed (Participants) | 75 | 75 | 31
percentage of participants | 68.0 | 54.7 | 87.1
Statistical Analysis 1: Comparison: Ibrutinib + Rituximab vs Placebo + Rituximab; Test type: Superiority; p = 0.1059, Cochran-Mantel-Haenszel — CMH chi squared test; Rate Ratio = 1.238, 95% CI 2-sided [0.955 to 1.603]

6. Secondary Outcome: Overall Survival (OS) - Kaplan Meier Landmark Estimates at Month 54
Description: OS, defined as the time from the date of randomization to the date of death from any cause. All deaths observed as the time of the analysis were considered as events. For participants who were not known to have died at the time of the analysis, OS data were censored at the date last known alive.
  As the median OS was not reached in any treatment arm at the time of the analysis, Kaplan Meier point estimates of the OS rate (that is, the estimated percentage of participants still surviving at Month 54) are presented.
Time Frame: Month 54 (median time on study: 49.7 months [Ibr+R and Pbo+R] and 57.9 months [Open-Label Ibr])
Population: Intent to Treat population: all randomized/enrolled participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ibrutinib + Rituximab | Placebo + Rituximab | Open-Label Substudy: Ibrutinib
Number analyzed (Participants) | 75 | 75 | 31
percentage of participants | 86.4 [73.7 to 93.3] | 84.2 [71.3 to 91.6] | 73.4 [53.7 to 85.7]
Statistical Analysis 1: Comparison: Ibrutinib + Rituximab vs Placebo + Rituximab; Data cutoff 18 December 2019; Test type: Superiority; p = 0.643, Log Rank — P-value is from unstratified log rank test; Hazard Ratio (HR) = 0.808, 95% CI 2-sided [0.328 to 1.99] — Hazard ratio is estimated using unstratified Cox regression model with treatment as the only covariate

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after the last dose of study drug. Median duration of treatment was 47.7 months for the Ibr+R arm, 15.5 months for the Pbo+R arm, and 40.7 months for the Open-Label Ibr arm.
Groups:
- Open-Label Substudy: Ibrutinib: Ibrutinib: 420 mg (3 capsules) orally administered daily beginning from Day 1 in Week 1 until progression, discontinuation due to toxicity or other reasons to discontinue treatment.
Arm/Group | Ibrutinib + Rituximab | Placebo + Rituximab | Open-Label Substudy: Ibrutinib
All-Cause Mortality (participants affected / at risk) | 9/75 | 10/75 | 8/31
Serious Adverse Events (participants affected / at risk) | 40/75 | 25/75 | 16/31
Other Adverse Events (participants affected / at risk) | 75/75 | 75/75 | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib + Rituximab (N=75) | Placebo + Rituximab (N=75) | Open-Label Substudy: Ibrutinib (N=31)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 8 | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 0 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Faecalith (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1
Death (General disorders) | 0 | 1 | 0 — Cause of death unknown
Fatigue (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1 | 0
Erysipelas (Infections and infestations) | 2 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 0 | 0
Hemianopia (Infections and infestations) | 0 | 0 | 1
Orchitis (Infections and infestations) | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 8 | 2 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0
Prostatic abscess (Infections and infestations) | 0 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 4 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 5 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Breast cancer metastatic (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Bing-Neel syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibrutinib + Rituximab (N=75) | Placebo + Rituximab (N=75) | Open-Label Substudy: Ibrutinib (N=31)
Anaemia (Blood and lymphatic system disorders) | 17 | 21 | 5
Increased tendency to bruise (Blood and lymphatic system disorders) | 9 | 2 | 8
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 12 | 7 | 9
Spontaneous haematoma (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 8 | 6
Atrial fibrillation (Cardiac disorders) | 11 | 1 | 0
Palpitations (Cardiac disorders) | 4 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 4
Cataract (Eye disorders) | 7 | 1 | 4
Diplopia (Eye disorders) | 0 | 0 | 2
Dry eye (Eye disorders) | 5 | 5 | 3
Eye irritation (Eye disorders) | 6 | 1 | 0
Lacrimation increased (Eye disorders) | 9 | 3 | 0
Photophobia (Eye disorders) | 6 | 2 | 0
Vision blurred (Eye disorders) | 7 | 2 | 4
Visual acuity reduced (Eye disorders) | 9 | 3 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 2
Vitreous floaters (Eye disorders) | 4 | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2 | 2
Constipation (Gastrointestinal disorders) | 9 | 9 | 5
Diarrhoea (Gastrointestinal disorders) | 23 | 11 | 14
Dry mouth (Gastrointestinal disorders) | 4 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 13 | 1 | 2
Gastritis (Gastrointestinal disorders) | 4 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 1 | 3
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 17 | 9 | 7
Stomatitis (Gastrointestinal disorders) | 4 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 8 | 0
Asthenia (General disorders) | 12 | 19 | 4
Chest pain (General disorders) | 4 | 0 | 0
Chills (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 13 | 18 | 5
Influenza like illness (General disorders) | 4 | 4 | 0
Oedema peripheral (General disorders) | 17 | 9 | 5
Pyrexia (General disorders) | 12 | 12 | 11
Bronchitis (Infections and infestations) | 11 | 5 | 3
Cellulitis (Infections and infestations) | 4 | 1 | 3
Conjunctivitis (Infections and infestations) | 4 | 3 | 4
Folliculitis (Infections and infestations) | 4 | 1 | 0
Herpes zoster (Infections and infestations) | 6 | 1 | 2
Influenza (Infections and infestations) | 10 | 5 | 2
Localised infection (Infections and infestations) | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 12 | 7 | 3
Oral herpes (Infections and infestations) | 6 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 2
Pneumonia (Infections and infestations) | 5 | 2 | 2
Respiratory tract infection (Infections and infestations) | 6 | 2 | 5
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 2
Rhinitis (Infections and infestations) | 4 | 1 | 2
Sinusitis (Infections and infestations) | 4 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 10 | 3 | 6
Urinary tract infection (Infections and infestations) | 11 | 0 | 3
Contusion (Injury, poisoning and procedural complications) | 7 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 7 | 3 | 3
Infusion related reaction (Injury, poisoning and procedural complications) | 32 | 43 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 5 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 7 | 3
Gout (Metabolism and nutrition disorders) | 4 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 2 | 0
Iron deficiency (Metabolism and nutrition disorders) | 4 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 9 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 7 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 | 9 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 6 | 5
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 0
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 35 | 0
Dizziness (Nervous system disorders) | 10 | 6 | 4
Headache (Nervous system disorders) | 13 | 17 | 7
Paraesthesia (Nervous system disorders) | 4 | 4 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 4 | 2
Sciatica (Nervous system disorders) | 6 | 0 | 3
Depression (Psychiatric disorders) | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 12 | 3 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 8 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 10 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 7 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 2
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Ecchymosis (Skin and subcutaneous tissue disorders) | 9 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 7 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 4 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 7 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 3 | 3
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 0 | 0
Hypertension (Vascular disorders) | 18 | 3 | 8
Hypotension (Vascular disorders) | 0 | 0 | 3
Blood Creatinine Increased (Investigations) | 5 | 0 | 0
Blood Uric Acid Increased (Investigations) | 4 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Institution/Investigator will not publish without Sponsor prior review and approval
2. Institution/Investigator will not publish until the earlier of (i) results of study are submitted for publication (ii) notification that submission of the multicenter results are no longer planned (iii) 18 months after study termination.

DOCUMENTS (2):
  • Study Protocol (2015-10-09): https://cdn.clinicaltrials.gov/large-docs/97/NCT02165397/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/97/NCT02165397/SAP_001.pdf